CLINICAL TRIAL: NCT00937339
Title: The Effects of Exercise and Whole Body Vibration Training on Bone Health, Physical Fitness, and Neuromotor Performance in Individuals With Chronic Stroke: A Randomized Controlled Trial.
Brief Title: Effects of Whole Body Vibration in People With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20090520002-01
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Stroke
Keywords: cerebrovascular accident; bone; muscle; vibration
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): The control group will perform the same exercises on the vibration platform, as in the experimental group. However, the vibration device will be turned off during the exercises.
  Interventions: Device: Exercise on the vibration platform with the device turned off
- Whole body vibration (Experimental): Subjects in the experimental group will undergo whole body vibration (1 session per day, 3 sessions per week) for 8 weeks. The vibration loading will be carried out using the Jet-Vibe System (Danil SMC Co., Ltd., Seoul, Korea). The vibration protocol used in this study will be 30Hz. While standing on the vibration platform, patients will be instructed to repeat the following set of light exercises: (1) light squatting,(2)deep squatting , (3) side-to-side weight-shift, (4) Forward and backward weight-shift, (5) forward lunge, (6) marching on the spot. The total duration of exposure of whole body vibration per session will be about 10 minutes.
  Interventions: Device: Whole body vibration therapy

INTERVENTIONS:
Device: Whole body vibration therapy — Experimental group: One session per day, 3 sessions per week, for consecutive 8 weeks. The total duration of whole body vibration therapy will be about 10 minutes per session.
  Other Names: Jet-Vibe System (Danil SMC Co., Ltd., Seoul, Korea)
  Arms: Whole body vibration
Device: Exercise on the vibration platform with the device turned off — Control group: One session per day, 3 sessions per week, for consecutive 8 weeks. The subjects will perform the same exercises on the vibration platform but no vibration will be applied.
  Other Names: Jet-Vibe System (Danil SMC Co., Ltd., Seoul, Korea)
  Arms: Control

SUMMARY:
The overall aim of the proposed study is to determine whether whole body vibration is beneficial in promoting bone health, physical fitness and neuromotor performance in patients with chronic stroke.

Subjects in the experimental group will undergo whole body vibration therapy (1 session per day, 3 sessions per week) for 8 weeks. The vibration frequency used in this study will be 30Hz. The total duration of exposure to vibration for the experimental group will be 10 minutes. While standing on the vibration platform, patients will be instructed to repeat the following set of light exercises: (1) light squatting,(2) deep squatting, (3) side-to-side weight-shift, (4) Forward and backward weight-shift, (5) forward lunge, (6) marching on the spot. The control exercise group, on the other hand, will perform the same exercise program on the platform, but no vibration will be given. The training will be conducted by a qualified personnel with physiotherapy background.

The outcome measurement will be performed 4 times: (1) immediately before the commencement of intervention, (2) immediately after termination of treatment, (3) at 1 month after termination of treatment. Each subject will be evaluated for bone markers, leg muscle strength, balance, spasticity, and walking ability.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of stroke more than 6 months
* medically stable
* able to understand verbal commands
* Abbreviated mental test score 6 or above
* age >18
* able to stand with or without aids for at least 1.5 minutes

Exclusion Criteria:

* neurological conditions other than stroke
* significant musculoskeletal conditions (e.g. amputations)
* metal implants in the lower extremity
* previous fracture of the lower extremity
* are currently taking bone resorption inhibitors or were taking the same before stroke.
* significant peripheral vascular disease
* vestibular disorders
* pregnancy
* Other serious illnesses that preclude the person from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Paretic knee concentric muscle strength | pre-test (week 0)
Paretic knee concentric muscle strength | Post-test (week 8)
Paretic knee concentric muscle strength | Follow-up (week 12)

SECONDARY OUTCOMES:
Non-paretic concentric knee muscle strength | Pre-test (week 0)
Non-paretic knee concentric muscle strength | Post-test (week 8)
Non-paretic knee concentric muscle strength | Follow-up (week 12)
Paretic knee eccentric muscle strength | pre-test (week 0)
Paretic knee eccentric muscle strength | Post-test (week 8)
Paretic knee eccentric muscle strength | WFollow-up (week 12)
Non-paretic knee eccentric muscle strength | Pre-test (week 0)
Non-paretic knee eccentric muscle strength | Post-test (week 8)
Non-paretic knee eccentric muscle strength | Follow-up (week 12)
Paretic knee isometric muscle strength | Pre-test (week 0)
Paretic knee isometric muscle strength | Post-test (week 8)
Paretic knee isometric muscle strength | Follow-up (week 12)
Non-paretic knee isometric muscle strength | Pre-test (week 0)
Non-paretic knee isometric muscle strength | Post-test (week 8)
Non-paretic knee isometric muscle strength | Follow-up (week 12)
Limit of stability test | Pre-test (week 0)
Limit of stability test | Post-test (week 8)
Limit of stability test | Follow-up (week 12)
Berg balance test | Pre-test (week 0)
Berg balance test | Post-test (week 12)
Berg balance test | Follow-up (week 12)
Activities-specific Balance Confidence Scale | Pre-test (week 0)
Activities-specific Balance Confidence Scale | Post-test (week 8)
Activities-specific Balance Confidence Scale | Follow-up (week 12)
Six Minute Walk Test | Pre-test (week 0)
Six Minute Walk Test | Post-test (week 8)
Six Minute Walk Test | Follow-up (week 12)
Self-selected gait velocity | Pre-test (week 0)
Self-selected gait velocity | post-test (week 8)
Self-selected gait velocity | Follow-up (week 12)
Bone formation marker level | pre-test (week 0)
Bone formation marker level | Post-test (week 8)
Bone resorption marker level | pre-test (week 0)
Bone formation marker level | Follow-up (week 12)
Bone resorption marker level | post-test (week 8)
Bone resorption marker level | Follow-up (week 12)
fall rate | 6 months after termination of treatment
Knee spasticity | Pre-test (week 0)
Knee spasticity | Post-test (week 8)
Knee spasticity | Follow-up (week 12)
Ankle spasticity | Pre-test (week 0)
Ankle spasticity | Post-test (week 8)
Ankle spasticity | Follow-up (week 12)
Level of satisfaction | Post-test (week 8)

CONTACTS AND LOCATIONS:
Overall Officials: Marco YC Pang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Hong Kong Polytechnic University, Hong Kong, China